CLINICAL TRIAL: NCT05808023
Title: Dose-dependent Individual FODMAPs (Mannitol and Fructans) Reintroduction in Patients With Irritable Bowel Syndrome
Brief Title: Dose-dependent FODMAP Reintroduction in IBS
Acronym: DORI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AZ Sint-Lucas Brugge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: S67424
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAP reintroduction; Fructans; Mannitol
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The patients will follow both reintroductions of fructans and mannitol in a randomized crossover way. The reintroduction periods are separated by a washout period of three days.
Who Masked: Participant
Masking Description: The patients will be blinded to both the dose and the tested powder sugar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol (Active Comparator): Mannitol belongs to the group of polyols within the FODMAPs.
  Interventions: Other: FODMAP powder reintroduction
- Fructans (Active Comparator): Fructans belong to the group of oligosaccharides, specifically the fructose-oligosaccharides (FOS), within the FODMAPs.
  Interventions: Other: FODMAP powder reintroduction

INTERVENTIONS:
Other: FODMAP powder reintroduction — The FODMAP powders will be reintroduced in three different doses, each for three consecutive days.

SUMMARY:
The aim of this study is to evaluate whether symptom recurrence, after successful FODMAP elimination, is dose-dependent in patients with IBS. The effect of a blinded reintroduction of FODMAP powders fructans and mannitol will be investigated in a crossover dose-escalation scheme for the identification of the eliciting dose in individual patients. The reintroduction of FODMAPs is performed after a successful elimination by the LFD.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Patients with irritable bowel syndrome according to Rome IV diagnostic criteria
4. Patients ages between 18 and 70 years old

Exclusion Criteria:

1. Participant has a history of any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years

1. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
2. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
3. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
4. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
5. Patients presenting with predominant symptoms of functional dyspepsia (FD) and of gastro-oesophageal reflux disease (GERD)
6. Patients following a diet interfering with the study diet in opinion of the investigator
7. Patients who already followed the low FODMAP diet under guidance of a trained dietitian without success.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose dependency | 18 months
  The study aims to determine the daily dose level of mannitol or fructans that induces symptom recurrence in IBS.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint Lucas, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No